CLINICAL TRIAL: NCT04703634
Title: The Effect of Ultrasound-guided Erector Spinae Block on Postoperative Analgesic Consumption in Patients Undergoing Nephrectomy. Prospective Randomized Single-center Study.
Brief Title: The Effect of Ultrasound-guided Erector Spinae Block on Postoperative in Patients Undergoing Nephrectomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Ayhan ŞAHİN, Asistant Prof, Namik Kemal University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2021-01-06; First posted 2021-01-11 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Nephrectomy
Keywords: erector spinae block; nephrectomy; ultrasound

STUDY DESIGN:
Intervention Model Description: It is a single centre, randomized, prospective method comparison study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- erector spinae group (Experimental): All blocks will be done under general anesthesia. Using a 6-10 MHz linear ultrasound (Esaote my-lab 6, Italy). With the ultrasonography device of our clinic, the side of the nephrectomy surgery will be performed with the position of the nephrectomy, and the position (lateral decubitus) is given to the patient. The thoracic 10th vertebra will be found under ultrasound guidance. After the T12 transverse protrusion is seen by sliding 3 cm laterally from the midline, 30 ml of 0.25% Bupivacaine will be injected under the erector spinae muscle above it.
  Interventions: Procedure: erector spinae block (ESP)
- placebo group (Placebo Comparator): No block transaction will be applied to this group. Only postoperative analgesia methods will be used for this group as specified in the protocol.
  Interventions: Procedure: erector spinae block (ESP)

INTERVENTIONS:
Procedure: erector spinae block (ESP) — Administration of local anesthetic under the erector spinae muscle just below the transverse process of the thoracic 12th vertebra

SUMMARY:
The main purpose of this study is to evaluate the postoperative effect of erector spinae block in patients undergoing nephrectomy that causes both visceral and somatic pain.

DETAILED DESCRIPTION:
After being informed and potential risks about the study, all patients have given written consent will undergo 24 hours screening for the analgesic effect of erector spinae block after nephrectomy. Patients meeting the criteria were randomly selected in double-blind manner 1:1 ratio to erector spiane block or not.

ELIGIBILITY:
Inclusion Criteria:

1. To undergo partial or total nephrectomy surgery
2. To be in ASA I-II classification
3. To be between the ages of 18-65.
4. Not having problems that prevent erector spinae block application such as local anesthetic drug allergy, infection at the injection site, and structural anomaly.
5. Being in good mental and psychological health
6. To accept to participate in the study.

Exclusion Criteria:

1. Being in ASA III or IV class with a high risk of anesthesia
2. Being outside the age range of 18-65
3. Having problems such as local anesthetic drug allergy, infection at the injection site, and structural anomaly prevents block application.
4. Not being mentally and psychologically healthy
5. Those who are allergic to the active substance, patients using antiepileptic drugs
6. Those with severe hepatic and renal failure
7. Those who have long-term use of nonsteroidal anti-inflammatory and opioid analgesic,
8. Those with diabetes and other neuropathic diseases
9. Patients who cannot use patient-controlled analgesia (PCA) device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | 24 hours
  Numerical Rating Scale (NRS) will be used for postoperative evaluation. NRS is a segmented digital version of the visual analog scale. Selecting an integer (0-10 integers) by a responder in (VAS). It is accepted as one dimensional-the measure of pain intensity in adults. The 11-point numerical scale ranges from "0" to "10," representing a pain ("no pain"). 10 ("as bad pain as you can imagine"), or ("the worst pain imaginable").

SECONDARY OUTCOMES:
Recovery analgesia | 24 hours
  Secondary outcome measures will be routine (paracetamol or tramadol PCA) or recovery. Analgesic use will be recorded within the first 24 hours.
postoperative nausea and vomiting | 24 hours
  The severity of nausea and vomiting 4-point scale (none, mild, moderate, and severe). As will be recorded by the nurses in the ward.

CONTACTS AND LOCATIONS:
Overall Officials: Ayhan ŞAHİN, Study Chair — Namık Kemal University Medicine Faculty
Locations (1):
- Namık Kemal University, Tekirdağ, Süleymanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be shared as much as the tasks described in the study. A meeting will be held at the end of the research, and the statistical data results will be shared. Dr. Ayhan Şahin is responsible.
Supporting Information: Study Protocol, SAP
Time Frame: starting after 6 months publication
Access Criteria: After publication, sharing will be made according to the journal criteria.